Official Title: GRAVITAS-309: A Phase 2/3 Study of Itacitinib and Corticosteroids as Initial

Treatment for Chronic Graft-Versus-Host Disease

NCT Number: NCT03584516

**Document Date**: Statistical Analysis Plan Amendment Version 1: 03 March 2022

## STATISTICAL ANALYSIS PLAN



# GRAVITAS-309: A Phase 2/3 Study of Itacitinib and Corticosteroids as Initial Treatment for Chronic Graft-Versus-Host Disease

| Sponsor: | Incyte Corporation 1801 Augustine Cut-Off Wilmington, DE 19803 |
|---|---|
| <b>Protocol Version:</b> | Protocol Amendment 8 dated 30 SEP 2021 |
| <b>CRF Approval Date:</b> | 13 OCT 2021 |
| SAP Version: | Amendment 1 |
| SAP Author: | , Biostatistics |
| Date of Plan: | 03 MAR 2022 |

This study is being conducted in compliance with good clinical practice, including the archiving of essential documents.

## TABLE OF CONTENTS

| TITLE I | PAGE | 1 |
|---------|-----------------------------------------------|----|
| TABLE | OF CONTENTS | 2 |
| LIST OF | F ABBREVIATIONS | 6 |
| 1. | INTRODUCTION | 8 |
| 1.1. | Preliminary Results From Part 1 | 8 |
| 1.2. | Rationale for Part 1 Expansion | 8 |
| 2. | STUDY INFORMATION, OBJECTIVES, AND ENDPOINTS | 9 |
| 2.1. | Protocol and Case Report Form Version | 9 |
| 2.2. | Study Objectives and Endpoints | 9 |
| 3. | STUDY DESIGN | 10 |
| 3.1. | Randomization | 11 |
| 3.1.1. | Part 1 | 11 |
| 3.1.2. | Part 1 Expansion | 11 |
| 3.2. | Control of Type I Error | 11 |
| 3.3. | Sample Size Considerations | 11 |
| 3.3.1. | Part 1 | 11 |
| 3.3.2. | Part 1 Expansion | 12 |
| 3.4. | Schedule of Assessments | 13 |
| 4. | DATA HANDLING DEFINITIONS AND CONVENTIONS | 13 |
| 4.1. | Scheduled Study Evaluations and Study Periods | 13 |
| 4.1.1. | Day 1 | 13 |
| 4.1.2. | Study Day | 13 |
| 4.1.3. | Baseline Value | 13 |
| 4.1.4. | Last Available Value | 14 |
| 4.1.5. | Handling of Missing and Incomplete Data | 14 |
| 4.2. | Variable Definitions | 14 |
| 4.2.1. | Body Mass Index | 14 |
| 4.2.2. | Body Surface Area | 14 |
| 4.2.3. | Prior and Concomitant Medication | 14 |
| 5. | STATISTICAL METHODOLOGY | 15 |
| 5.1. | General Methodology | 15 |

| 5.2. | Treatment Groups | 15 |
|---|---|---|
| 5.2.1. | Part 1 | 15 |
| 5.2.2. | Part 1 Expansion | 15 |
| 5.3. | Analysis Populations | 15 |
| 6. | BASELINE, EXPOSURE, AND DISPOSITION VARIABLES AND ANALYSES | 16 |
| 6.1. | Baseline Demographics, Physical Characteristics, and Disease History | 16 |
| 6.1.1. | Demographics and Baseline Characteristics | 16 |
| 6.1.2. | Disease History for Chronic Graft-Versus-Host Disease | 16 |
| 6.1.3. | Medical History | 16 |
| 6.1.4. | Primary Hematologic Disease and Transplant Characteristics | 16 |
| 6.2. | Disposition of Participants | 16 |
| 6.3. | Protocol Deviations | 17 |
| 6.4. | Exposure | 17 |
| 6.5. | Study Drug Compliance | 18 |
| 6.6. | Prior and Concomitant Medication | 18 |
| 7. | EFFICACY | 19 |
| 7.1. | General Considerations | 19 |
| 7.2. | Primary Analysis | 19 |
| 7.3. | Analyses of the Secondary Efficacy Parameters | 19 |
| 7.3.1. | Response Rate | 19 |
| 7.3.2. | Time to Response | 20 |
| 7.3.3. | Duration of Response | 20 |
| 7.3.4. | Best Overall Response | 21 |
| 7.3.5. | Overall Survival | 21 |
| 7.3.6. | Nonrelapse Mortality Rate | 21 |
| 7.3.7. | Relapse Rate of Malignant and Nonmalignant Hematologic Diseases | 21 |
| 7.3.8. | Time to Primary Hematologic Disease Relapse | 21 |
| 7.3.9. | Other Efficacy Analyses | 22 |
| 8. | PHARMACOKINETIC ANALYSES | 22 |
| 8.1. | Pharmacokinetic Analyses | 22 |
| | | 22 |
| 9. | SAFETY AND TOLERABILITY | 23 |

| 9.1. | General Considerations | 23 |
|---|---|---|
| 9.2. | Adverse Events | 23 |
| 9.2.1. | Adverse Event Definitions | 23 |
| 9.2.2. | Dose-Limiting Toxicities | 24 |
| 9.2.3. | Adverse Event Summaries | 25 |
| 9.2.4. | Clinically Notable Adverse Events Based on Customized MedDRA Queries | 27 |
| 9.3. | Analyses for the Data Monitoring Committee | 27 |
| 9.4. | Clinical Laboratory Tests | 27 |
| 9.5. | Vital Signs | 27 |
| 9.6. | Electrocardiograms | 28 |
| 10. | INTERIM ANALYSES | 28 |
| 11. | CHANGES AND MODIFICATIONS TO THE ANALYSIS PLAN | 28 |
| 11.1. | Changes to Protocol-Defined Analyses | 28 |
| 11.2. | Changes to the Statistical Analysis Plan | 28 |
| 12. | REFERENCES | 29 |
| APPENDI | X A. PLANNED TABLES AND LISTINGS | 30 |
| APPENDI | X B. CLINICALLY NOTABLE HEMATOLOGIC EVENTS | 34 |
| APPENDI | X C. HEMATOLOGIC INFECTION EVENTS | 35 |
| APPENDI | X D. HYPERLIPIDEMIA EVENTS | 36 |
| APPENDI | X E. QT PROLONGATION EVENTS | 38 |
| APPENDI | X F. THROMBOEMBOLIC EVENTS | 39 |
| APPENDI | X G. PLANNED TABLES AND FIGURES FOR PHARMACOKINETIC AND PHARMACOKINETIC/PHARMACODYNAMIC ANALYSIS | 45 |
| | LIST OF TABLES | |
| Table 1: | Objectives and Endpoints, Part 1 and Part 1 Expansion | 9 |
| Table 2: | Treatment Groups and Dose Levels and Schedules | 11 |
| Table 3: | Bayesian Posterior Probability to Demonstrate That There Is a Clinically Meaningful Difference Between Any Itacitinib Group and the Corticosteroids-Only Group | 12 |
| Table 4: | Populations for Analysis | |
| Table 5: | Definitions of Dose-Limiting Toxicity | 24 |
| Table 6: | | |

| Incyte Corporation INCB 39110-309 Statistical Analysis Plan Am 1 | | Page 5 of 45<br>03 MAR 2022 |
|---|---|---|
| Table 7: | Criteria for Vital Sign Abnormalities | 27 |
| Table 8: | Statistical Analysis Plan Versions | 28 |

## LIST OF ABBREVIATIONS

| Abbreviation | Term |
|---|---|
| AE | adverse event |
| aGVHD | acute graft-versus-host disease |
| AUC | area under the plasma or serum concentration-time curve |
| AUC <sub>0-t</sub> | area under the plasma or serum concentration-time curve from time $= 0$ to the last measurable concentration at time $= t$ |
| BID | twice daily |
| BMI | body mass index |
| BOR | best overall response |
| BSA | body surface area |
| cGVHD | chronic graft-versus-host disease |
| CI | confidence interval |
| Cl/F | apparent oral dose clearance |
| $C_{max}$ | maximum observed plasma or serum concentration |
| C <sub>min</sub> | minimum observed plasma or serum concentration |
| CMV | cytomegalovirus |
| CR | complete response |
| CRF | case report form |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DLT | dose-limiting toxicity |
| DMC | Data Monitoring Committee |
| DoR | duration of response |
| EBV | Epstein-Barr virus |
| eCRF | electronic case report form |
| GVHD | graft-versus-host disease |
| ITT | intent-to-treat |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MQ | MedDRA query |
| NCI | National Cancer Institute |
| NIH | National Institutes of Health |
| NRM | nonrelapse mortality |
| ORR | objective response rate |
| OS | overall survival |
| PK | pharmacokinetic |
| PR | partial response |
| PT | preferred term |

| Abbreviation | Term |
|------------------|----------------------------------|
| QD | once daily |
| SAP | Statistical Analysis Plan |
| SOC | system organ class |
| TEAE | treatment-emergent adverse event |
| $T_{\text{max}}$ | time to maximum concentration |
| WHO | World Health Organization |

#### 1. INTRODUCTION

This is a 2-part, Phase 2/3 study of itacitinib or placebo in combination with corticosteroids as initial treatment for cGVHD. Part 1 is a run-in that will employ a randomized, open-label, parallel-cohort design with the primary objective to assess the safety and tolerability of itacitinib in combination with corticosteroids in order to identify the appropriate dose of itacitinib in combination with corticosteroids as initial treatment for moderate or severe cGVHD. A total of 20 participants with moderate or severe cGVHD will be randomized 1:1 to itacitinib 200 mg QD plus corticosteroids or 300 mg QD plus corticosteroids.

Part 1 expansion is a Phase 2 with an initial safety run-in that will employ a randomized, open-label, parallel-cohort design with the primary objective to assess the safety and preliminary efficacy of itacitinib in combination with corticosteroids compared with corticosteroids monotherapy and identify the appropriate dosing/schedule of itacitinib in combination with corticosteroids as initial treatment for cGVHD for Part 2. A total of up to 140 participants (35 per treatment group) with moderate or severe cGVHD will be randomized 1:1 to 1 of 4 treatment groups: itacitinib 300 mg QD plus corticosteroids (Treatment Group A), itacitinib 400 mg QD plus corticosteroids (Treatment Group B), itacitinib 300 mg BID plus corticosteroids (Treatment Group C), or corticosteroids monotherapy (Treatment Group D). Randomization will be stratified by cGVHD risk status (moderate vs severe). Treatment Groups B and C will have an initial safety run-in of 10 participants to determine safety and tolerability of the dose before expansion. Participants enrolled in the safety run-in will be monitored continuously. Treatment Group C was discontinued as of Amendment 8, and participants in that treatment group who were ongoing were allowed to reduce to 400 mg QD plus corticosteroids.

The purpose of the original version of the SAP was to provide details of the statistical analyses that have been outlined in Part 1 of the Protocol.

The purpose of Amendment 1 is to provide details of the statistical analyses that have been outlined in Part 1 expansion of Protocol Amendment 8.

## 1.1. Preliminary Results From Part 1

Preliminary data from Part 1 were reviewed by an independent DMC, and the summary data are presented in the Protocol. The DMC recommended that 300 mg QD be chosen as the Part 2 dose of itacitinib as no differences emerged between the doses with respect to toxicity.

## **1.2.** Rationale for Part 1 Expansion

Additional dosing regimens of itacitinib were selected for evaluation in combination with corticosteroids in an expansion to Part 1 of the study, and the underlying rationale is presented in the Protocol.

## 2. STUDY INFORMATION, OBJECTIVES, AND ENDPOINTS

## 2.1. Protocol and Case Report Form Version

This amendment of the SAP is based on INCB 39110-309 Protocol Amendment 8 dated 30 SEP 2021 and CRFs approved 13 OCT 2021.

## 2.2. Study Objectives and Endpoints

Study objectives and endpoints for Part 1 and Part 1 expansion are shown in Table 1.

Table 1: Objectives and Endpoints, Part 1 and Part 1 Expansion

| Objectives | Endpoints |
|---|---|
| Primary | |
| To identify an appropriate dose of itacitinib in combination with corticosteroids as initial treatment for moderate or severe cGVHD. | Part 1: DLT data through Day 28 and additional data from clinical safety and laboratory assessments. Part 1 expansion: Incidence and severity of adverse events, across treatment cohorts. |
| Key Secondary (for Part 1 Expansion) | da verse e venis, de ress de danere e enercia |
| To evaluate preliminary activity across treatment cohorts with respect to response rate at Month 3 and Month 6. | Response rate at Month 3 and Month 6, defined as the proportion of participants who demonstrate a CR or PR at each timepoint. |
| Secondary | |
| To evaluate the PK of itacitinib when administered in combination with corticosteroids in the study population. | C <sub>max</sub> , C <sub>min</sub> , T <sub>max</sub> , AUC <sub>0-t</sub> , and Cl/F. |
| To estimate efficacy outcomes for each treatment cohort. | Part 1: Response rate at Month 3, 6, and 12. Part 1 expansion: Response rate at Month 12. Response rate is defined as the proportion of participants who demonstrate either a CR or PR at each timepoint. |
| | Time to response, defined as the interval between randomization and first response. |
| | DoR, defined as the interval between first response and cGVHD progression, death, or initiation of new systemic cGVHD therapy. |
| | OS, defined as the interval between the date of randomization and the date of death due to any cause. |
| | NRM, defined as the proportion of participants who died due to causes other than a relapse of their primary hematologic disease. |
| | Proportion of participants with ≥ 50% reduction in daily corticosteroid dose at Day 180. |

Table 1: Objectives and Endpoints, Part 1 and Part 1 Expansion (Continued)

| Objectives | Endpoints |
|---|---|
| To estimate efficacy outcomes for each treatment cohort (continued). | Proportion of participants successfully tapered off all corticosteroids at Day 180. |
| | Relapse rate of malignant and nonmalignant hematologic diseases, defined as the proportion of participants whose underlying disease relapses. |
| | Time to primary hematologic disease relapse, defined as the interval between the date of randomization and the date of relapse. |
| | randomization and the date of relapse. |

### 3. STUDY DESIGN

Part 1 is a run-in that will employ a randomized, open-label, parallel-cohort design to assess the safety and tolerability of itacitinib in combination with corticosteroids in order to identify the appropriate dose level for initial treatment of moderate or severe cGVHD. A total of 20 participants with moderate or severe cGVHD will be randomized 1:1 to itacitinib 200 mg QD plus corticosteroids or 300 mg QD plus corticosteroids. Itacitinib treatment will continue until treatment failure (cGVHD progression, death, or initiation of new systemic cGVHD therapy), unacceptable toxicity, or withdrawal of consent, for a maximum of 36 months. Participants may remain on study for a total of 37 months, including the treatment period, safety follow-up, and post-treatment GVHD follow-up, unless death or withdrawal of consent occurs earlier.

Chronic GVHD staging and grading will be assessed using NIH consensus guidelines (Jagasia et al 2015, Lee et al 2015); safety and tolerability will be assessed as per NCI CTCAE v4.03.

An analysis to determine the dose for further study will be performed once the 20th evaluable participant completes 28 days of study treatment. An external DMC will review data from this analysis and provide a recommendation on an appropriate dose for Part 2.

In Part 1, any participant who withdraws from treatment before the completion of the 28-day observation period for any reason other than a DLT (eg, not evaluable for DLT) may be replaced to ensure a minimum number of evaluable participants.

Part 1 expansion is a Phase 2 with an initial safety run-in that will employ a randomized, open-label, parallel-cohort design with the primary objective to assess the safety and preliminary efficacy of itacitinib in combination with corticosteroids compared with corticosteroids monotherapy and identify the appropriate dosing/schedule of itacitinib in combination with corticosteroids as initial treatment for cGVHD for Part 2. A total of up to 140 participants (35 per treatment group) with moderate or severe cGVHD will be randomized 1:1 to 1 of 4 treatment groups (see Table 2): itacitinib 300 mg QD plus corticosteroids (Treatment Group A), itacitinib 400 mg QD plus corticosteroids (Treatment Group B), itacitinib 300 mg BID plus corticosteroids (Treatment Group C), or corticosteroids monotherapy (Treatment Group D).

**Table 2:** Treatment Groups and Dose Levels and Schedules

| Treatment<br>Group | Dose Level and Schedule |
|---|---|
| A | Itacitinib 300 mg QD plus corticosteroids |
| В | Itacitinib 400 mg QD plus corticosteroids |
| С | Itacitinib 300 mg BID plus corticosteroids; may be decreased to 200 mg BID if a boundary is reached during safety run-in. This treatment group was discontinued due to concern of a potential increase in relapse rate. Participants in this treatment group who were ongoing were allowed to reduce to 400 mg QD plus corticosteroids. |
| D | Corticosteroids monotherapy |

## 3.1. Randomization

#### 3.1.1. Part 1

A total of 20 participants with moderate or severe cGVHD will be randomized 1:1 to itacitinib 200 mg QD plus corticosteroids or 300 mg QD plus corticosteroids.

## 3.1.2. Part 1 Expansion

A total of up to 140 participants (35 per treatment group) with moderate or severe cGVHD will be randomized 1:1 to 1 of 4 treatment groups: itacitinib 300 mg QD plus corticosteroids (Treatment Group A), itacitinib 400 mg QD plus corticosteroids (Treatment Group B), itacitinib 300 mg BID plus corticosteroids (Treatment Group C), or corticosteroids monotherapy (Treatment Group D).

Randomization will be stratified by cGVHD risk status (moderate vs severe). Treatment Groups B and C will have an initial safety run-in of 10 participants to determine safety and tolerability of the dose before expanding (see definition of DLT in Section 6.1.1.3 of the Protocol). Participants enrolled in the safety run-in will be monitored continuously using the Bayesian approach. Treatment Group C was discontinued as of Amendment 8, and participants in that treatment group who were ongoing were allowed to reduce to 400 mg QD plus corticosteroids.

## 3.2. Control of Type I Error

No formal statistical tests will be performed in Part 1 and Part 1 expansion. All CIs will be 95%.

## 3.3. Sample Size Considerations

#### 3.3.1. Part 1

In Part 1, approximately 20 participants will be enrolled to achieve 10 randomly assigned participants in each of the 2 dose groups of itacitinib in order to identify an optimal dose for further study. This sample size was chosen based on typical Phase 1 studies employing a 3 + 3 design that enroll up to 9 participants in order to identify recommended Phase 2 doses. A sample size of 20 participants (10 per treatment group) allows for concurrent enrollment at 2 dose levels

that have been previously characterized in other disease settings and is expected to enable the clinical characterization of study treatment across 2 treatment cohorts. No formal statistical comparison will be performed between treatment groups.

## 3.3.2. Part 1 Expansion

Sample size in Part 1 expansion is based on clinical feasibility and consideration. No hypothesis test is planned for efficacy. Up to 35 participants will be enrolled into each treatment group. The toxicity of itacitinib will be monitored continuously for Treatment Groups B and C using a Bayesian approach. A total of up to 140 participants will be enrolled into Part 1 expansion of the study. Regarding the key secondary endpoint, Month 6 response rate, a table of Bayesian posterior probabilities and related descriptions are provided below. This posterior probability may be used to support decision-making on itacitinib dosing/schedule for Part 2, including decisions made by the DMC

Table 3 presents Bayesian posterior probability of demonstrating a clinically meaningful treatment difference in Month 6 response rate between any itacitinib group and the corticosteroids-only group under various response rates at the end of the expansion.

Table 3: Bayesian Posterior Probability to Demonstrate That There Is a Clinically Meaningful Difference Between Any Itacitinib Group and the Corticosteroids-Only Group

| Responders in an Itacitinib Group | Responders in Corticosteroids-Only Group (out of 35) | | | | |
|---|---|---|---|---|---|
| (out of 35) | 18 | 19 | 20 | 21 | 22 |
| 25 | 64.3% | 54.8% | 45.0% | 35.3% | 26.4% |
| 26 | 73.1% | 64.4% | 54.9% | 44.8% | 35.0% |
| 27 | 80.9% | 73.4% | 64.7% | 54.9% | 44.7% |
| 28 | 87.2% | 81.3% | 73.9% | 65.0% | 55.0% |
| 29 | 92.1% | 87.7% | 81.9% | 74.4% | 65.3% |
| 30 | 95.5% | 92.6% | 88.4% | 82.6% | 75.0% |

Note: With a binomial likelihood, binomial (n, p) with s number of responders out of n participants, and a beta prior, Beta (a, b), the posterior is calculated as Beta(a+s, b+n-s).

#### Interpretation:



#### 3.4. Schedule of Assessments

Refer to Protocol Amendment 8 dated 30 SEP 2021 for a full description of all study procedures and assessment schedules for this study.

### 4. DATA HANDLING DEFINITIONS AND CONVENTIONS

## 4.1. Scheduled Study Evaluations and Study Periods

## 4.1.1. Day 1

Day 1 is the date that the first dose of itacitinib is administered to the participants. For the corticosteroids-only group, Day 1 will be defined as the first nonmissing dose day.

## **4.1.2. Study Day**

If a visit/reporting date is on or after Day 1, then the study day at the visit/reporting date will be calculated as

Day # = (visit/reporting date - Day 1 date + 1).

If the visit/reporting date is before Day 1, then the study day at the visit/reporting date will be calculated as

Day # = (visit/reporting date - Day 1 date).

A study day of -1 indicates 1 day before Day 1.

#### 4.1.3. Baseline Value

Baseline is the last nonmissing measurement obtained before the first administration of study treatment (eg, itacitinib with corticosteroids or corticosteroids only). When itacitinib and corticosteroids are started on different days, then the rules mentioned in Section 4.1.1 will be followed.

When scheduled assessments and unscheduled assessments occur on the same day, and time of the assessment or time of first dose is not available, use the following convention to determine baseline:

- If both a scheduled and an unscheduled visit are available on the day of the first dose and the time is missing, use the scheduled assessment as baseline.
- If all scheduled assessments are missing on the day of the first dose and an unscheduled assessment is available, use the unscheduled assessment as baseline.

#### 4.1.4. Last Available Value

The last available value is the last nonmissing measurement obtained after starting the study treatment.

## 4.1.5. Handling of Missing and Incomplete Data

Missing observations will be handled for specific endpoints as detailed in the sections addressing each analysis.

#### 4.2. Variable Definitions

## 4.2.1. Body Mass Index

Body mass index will be calculated as follows:

BMI 
$$(kg/m^2) = [weight (kg)] / [height (m)]^2$$

## 4.2.2. Body Surface Area

Body surface area will be calculated based on the Mosteller (1987) formula as follows:

Sites will also record the BSA calculated per institutional standards.

#### 4.2.3. Prior and Concomitant Medication

Prior medication is defined as any nonstudy medication started before the first dose of itacitinib or corticosteroids for participants on corticosteroids only in the Part 1 expansion.

Concomitant medication is defined as any nonstudy medication that is started accordingly:

- Before the date of first administration of itacitinib or corticosteroids only and is ongoing throughout the study or ends on/after the date of first itacitinib or corticosteroid administration.
- On/after the date of first administration of itacitinib or corticosteroids only and is ongoing or ends during the course of itacitinib or corticosteroid treatment.

A prior medication could also be classified as "both prior and concomitant medication" if the end date is on or after the first dose of itacitinib or corticosteroids only. Since corticosteroids are part of the study medication, they will not appear in the list of prior and concomitant medications unless prescribed for an indication other than GVHD. In the listing, it will be indicated whether a medication is prior only, concomitant only, or both prior and concomitant.

For the purposes of analysis, all medications will be considered concomitant medications unless the medications can unequivocally be defined as not concomitant.

### 5. STATISTICAL METHODOLOGY

## 5.1. General Methodology

Unless otherwise noted, SAS® software (SAS Institute Inc, Cary, NC; v9.4 or later) will be used for the generation of all tables, graphs, and statistical analyses. Descriptive summaries for continuous variables will include, but not be limited to, the number of observations, mean, standard deviation, median, minimum, and maximum. Descriptive summaries for categorical variables will include the number and percentage of participants in each category.

## **5.2.** Treatment Groups

#### 5.2.1. Part 1

A total of 20 participants with moderate or severe cGVHD will be randomized 1:1 to itacitinib 200 mg QD plus corticosteroids or itacitinib 300 mg QD plus corticosteroids.

## 5.2.2. Part 1 Expansion

A total of up to 140 participants (35 per treatment group) with moderate or severe cGVHD will be randomized 1:1 to 1 of 4 treatment groups: itacitinib 300 mg QD plus corticosteroids (Treatment Group A), itacitinib 400 mg QD plus corticosteroids (Treatment Group B), itacitinib 300 mg BID plus corticosteroids (Treatment Group C), or corticosteroids monotherapy (Treatment Group D).

## 5.3. Analysis Populations

The populations that will be included in study-related analyses are described in Table 4.

**Table 4: Populations for Analysis** 

| Population | Description |
|---|---|
| ITT | All randomized participants |
| Safety | All enrolled/randomized participants who received at least 1 dose of study drug and/or reference therapy. Treatment groups for this population will be determined according to the actual treatment the participant received regardless of assigned study drug treatment. |
| Safety run-in | All participants enrolled in the safety run-in portion of the study who received at least 1 dose of study drug and/or reference therapy. Treatment groups for this population will be determined according to the treatment assignment on Day 1 regardless of the actual study drug the participant might take during their continued participation in the study. |
| PK evaluable | All participants who received at least 1 dose of study drug and/or reference therapy and provided at least 1 postdose plasma sample (1 PK measurement). The study pharmacokineticist will review data listings of study drug administration and sample records to identify participants to be excluded from analyses of PK data. |

## 6. BASELINE, EXPOSURE, AND DISPOSITION VARIABLES AND ANALYSES

Appendix A provides a list of planned tables, figures, and listings.

## 6.1. Baseline Demographics, Physical Characteristics, and Disease History

Demographic and baseline characteristics, disease history, and prior therapy will be summarized for the safety run-in and Part 1 expansion populations and listed.

## **6.1.1.** Demographics and Baseline Characteristics

The following demographic and baseline characteristics will be summarized for the safety run-in population and Part 1 expansion: age, sex, race, ethnicity, weight (by sex), height, BMI, BSA, and Karnofsky performance status.

### 6.1.2. Disease History for Chronic Graft-Versus-Host Disease

Baseline cGVHD staging and grading, time since diagnosis of cGVHD, organs involved, aGVHD (yes/no) and grade, conditioning and prophylaxis therapy, donor type, and other details related to the disease under study and transplant will be summarized at baseline. Day 1 assessment will be used to determine baseline organ involvement.

Time since cGVHD diagnosis will be calculated as:

Time since diagnosis (years) = (Day 1 date – date of diagnosis + 1) / 365.25.

## **6.1.3.** Medical History

For participants in the safety run-in population and participants in the Part 1 expansion, medical history will be summarized by assigned treatment group. This summation will include the number and percentage of participants for each body system/organ class as documented on the eCRF.

### 6.1.4. Primary Hematologic Disease and Transplant Characteristics

Summary will include disease-targeted medical and treatment history such as participant's primary hematologic disease, including diagnosis, prior therapy, disease stage at the time of transplantation, disease risk index, and details regarding allogeneic hematopoietic stem cell transplantation; prior and current GVHD prophylaxis; history of aGVHD; and current cGVHD staging information.

Cancer history and underlying hematologic disease will also be summarized.

## **6.2.** Disposition of Participants

The number and percentage of participants who were randomized, treated, completed treatment, discontinued study treatment with a primary reason for discontinuation, and withdrew from the study with a primary reason for withdrawal will be summarized for the safety run-in population and the Part 1 expansion population.

#### 6.3. Protocol Deviations

Protocol deviations recorded on the eCRF will be summarized and presented in the participant data listings.

## 6.4. Exposure

For participants in the safety run-in population and participants in the Part 1 expansion, exposure to itacitinib and corticosteroids will be summarized descriptively as follows.

#### • Duration of treatment with itacitinib:

The exposure start date is when trt = itacitinib and exposure timepoint = first dose; when a participant does not have first dose record (but has other timepoints) as the exposure timepoint, exposure start date should be when trt = itacitinib and dose is not missing.

Duration of treatment (days) = Date of last dose of itacitinib – Date of first dose of itacitinib + 1.

## • Average daily dose of itacitinib:

Average daily dose (mg/day) = Total actual itacitinib dose taken (mg) / Duration of treatment with itacitinib (days).

#### • Dose modifications of itacitinib:

Numbers of participants who had itacitinib dose reduction and/or interruption will be summarized. Separate summaries will be generated for participants with dose change due to dose tapering (change of dose due to efficacy of treatment) and participants with dose change due to other reasons (potential safety concerns).

#### Duration of treatment with corticosteroids:

For corticosteroids, the first exposure start date is when the dose is not missing.

Duration of treatment (days) = Date of last dose of corticosteroid – Date of first dose of corticosteroid + 1.

If a participant is being treated with a corticosteroid prior to Day 1, study Day 1 will be used if no other data are available to conform to the definition provided in Section 4.1.1. If a participant is prescribed a corticosteroid for a flare during the course of the study, duration of treatment will be adjusted to account for the break in treatment between completing taper and starting of a short pulse for a flare.

### • Average daily dose of corticosteroids:

Average daily dose (mg/day) = Total actual corticosteroid dose taken (mg) / Duration of treatment with corticosteroids (days).

Daily dose will account for how the doses are prescribed (eg, BID is converted to twice daily).

## Reduction in daily dose of corticosteroids and successful tapering of corticosteroids

Numbers of participants who had dose reduction and/or interruption of corticosteroids will be summarized as follows:

- Summary of number of participants with ≥ 50% reduction in daily corticosteroid dose at Day 180
- Summary of participants successfully tapered off all corticosteroids at Day 180
- Summary of number of participants with  $\geq 50\%$  reduction in daily corticosteroid dose by (4-week) time interval up to Month 6
- Summary of participants successfully tapered off all corticosteroids by (4-week) time interval up to Month 6

Participants will be considered as having a competing risk at the time of cGVHD progression or start of a new systemic therapy for cGVHD, relapse of the underlying hematologic disease, or death.

Sensitivity analyses may be performed for participants who had their corticosteroid dose increased during the corticosteroid taper period for a non-GVHD medical condition.

## **6.5.** Study Drug Compliance

For participants in the safety run-in population and participants in the Part 1 expansion, overall compliance (%) for the study treatment will be calculated for all participants as follows:

Compliance (%) =  $100 \times [\text{total dose actually taken}] / [\text{total prescribed dose}].$ 

The total prescribed dose is defined as the sum of the doses prescribed by the investigator accounting for dose modifications.

### 6.6. Prior and Concomitant Medication

For participants in the safety run-in population and participants in Part 1 expansion, prior medications and concomitant medications will be coded using the WHO Drug Dictionary and summarized by WHO drug class and WHO drug term. Results will be summarized as number and percentage of participants with prior and concomitant medications by PT and WHO drug class.

#### 7. EFFICACY

Appendix A provides a list of planned tables, figures, and listings.

### 7.1. General Considerations

In Part 1, all efficacy analyses will be performed using the safety run-in population. In Part 1 Expansion, all efficacy analyses will be performed using the safety population.

If there are not sufficient data for meaningful statistical inference, the planned analysis will not be performed, and only related summary statistics and/or listings will be provided.

In all efficacy analyses, initiation of new systemic anti-GVHD therapy includes 4 scenarios:

- 1. Initiation of new anti-GVHD therapy including a higher dose of corticosteroid than that used at Day 1.
- 2. The need for a second dose increase in corticosteroids.
- 3. A dose increase in corticosteroids that is not tapered back to the previous dose of corticosteroids within 6 weeks ( $\pm$  2 days) of the increase.
- 4. Reintroduction of systemic corticosteroids that occurs after complete taper of corticosteroids due to response.

No formal statistical tests will be performed.

## 7.2. Primary Analysis

In Part 1, the primary objective is to identify an appropriate dose of itacitinib (200 mg QD or 300 mg QD) in combination with corticosteroids as initial treatment for moderate or severe cGVHD. The DLT data through Day 28 and additional data from clinical safety and laboratory assessments will be used as primary endpoints for this analysis.

In Part 1 Expansion, the primary objective is to identify an appropriate dose of itacitinib (300 mg QD, 400 mg QD, or 300 mg BID) in combination with corticosteroids as initial treatment for moderate or severe cGVHD. The selection of the dose is primarily based on the incidence and severity of AEs across treatment cohorts and will be supported by cGVHD response data (refer to Section 10.1.2 of the Protocol).

## 7.3. Analyses of the Secondary Efficacy Parameters

#### 7.3.1. Response Rate

Response rate at 3, 6, and 12 months (Days 90, 180, and 365) is defined as the proportion of participants who achieved a response (CR or PR) at each of these timepoints based on an ITT population.

A participant will not be considered a responder for the analysis of ORR at 3, 6, and 12 months if any of the following events occurred at or prior to the response assessment at the predefined timepoint:

• cGVHD progression per NIH response criteria or initiation of a new systemic therapy for cGVHD

- Evidence of progression of the underlying hematologic disease
- Withdrawal from the study
- Death
- Response assessment missing (not performed) at the predefined timepoint

The proportion of responders will be estimated with 95% CIs. Confidence intervals will be calculated based on the exact method for binomial distributions. Summary statistics will be provided.

Additional analyses may be performed based on evaluable subsets. An evaluable population will also be considered with participants who have completed 3, 6, or 12 months of follow-up as of the cutoff date or discontinued earlier because of new cGVHD progression. Presentations of ORR at Month 3 and Month 6 will include a footnote explaining what "evaluable" means (ie, participants who had at least 3 or 6 months of follow-up as of the cutoff date or discontinued earlier).

Summary statistics and 95% CI will be provided by cohort. The primary comparisons in Part 1 expansion will involve only the 2 itacitinib groups (Treatment Groups A and B) and the corticosteroids-only group (Treatment Group D) as a result of Protocol Amendment 8, in which Treatment Group C (300 mg BID + corticosteroids) was discontinued. Data from Treatment Group C will be presented only as summary statistics and will not be subjected to any statistical comparison.

Pairwise Cochran-Mantel-Haenszel tests will be conducted for Month 6 response rate for each of the 2 itacitinib groups (Treatment Groups A and B) and the corticosteroids-only group (Treatment Group D) as an exploratory analysis.

The secondary endpoints discussed below will be summarized by Treatment Groups A, B, and D using the ITT population for efficacy-related endpoints and all groups for safety-related endpoints.

#### 7.3.2. Time to Response

Time to response is defined as the interval from randomization to first response (CR or PR) before initiation of new therapy. In the time to response analysis, participants without a response after randomization will be censored at either study withdrawal, initiation of new systemic anti-GVHD therapy, death, relapse, or last response assessment prior to or on the cutoff date, whichever is earliest. Time to response will be summarized for participants who achieve a response using the Kaplan-Meier method. Median time to response and a 95% CI will be estimated.

### 7.3.3. **Duration of Response**

Duration of response is defined as the interval between the date of initial documentation of response (CR or PR) and the date of cGVHD progression per NIH response criteria, initiation of new systemic cGVHD therapy, or death. Participants experiencing relapse of underlying hematologic relapse will be censored at the date of relapse.

Duration of response will be summarized for participants who achieve a response. Duration of response will be assessed using the Kaplan-Meier method for participants who achieve a response. Median duration and a 95% CI will be estimated. Participants who are still responding at the time of database lock or discontinuation will be right-censored at the time of last valid response assessment.

#### 7.3.4. Best Overall Response

Best overall response for each participant is defined as best response during the course of the study (best in the categories of CR or PR), including responses at unscheduled visits. Participants without a BOR (ie, participants not achieving a response of either CR or PR) in the treatment phase will be considered as nonresponders for BOR in the responder analysis. Number and percentage of participants in each best response category will be tabulated by treatment group.

#### 7.3.5. Overall Survival

Overall survival is defined as the interval between the date of randomization and the date of death due to any cause. Date of death will be determined using the Death Report, the Survival Follow-Up, and the Subject Status CRFs. The Kaplan-Meier method will be used to estimate the survival time distribution and the median survival, if it is applicable. Participants with no observed death or loss to follow-up will be treated as censored at their last date known to be alive. The 95% CI will be calculated using Brookmeyer and Crowley's method (1982). Summary statistics will be provided.

## 7.3.6. Nonrelapse Mortality Rate

Nonrelapse mortality is defined as the time from date of randomization to date of death not preceded by underlying disease relapse/recurrence. Underlying disease relapse/recurrence is considered a competing event. If a participant is not known to have died or experienced the competing event, then NRM will be censored at the latest date the participant was known to be event-free (on or before the cutoff date). Cumulative incidence of NRM and derived probabilities at Months 3, 6, and 12 will be estimated, considering underlying disease relapse/recurrence as a competing event.

## 7.3.7. Relapse Rate of Malignant and Nonmalignant Hematologic Diseases

Relapse rate of malignant and nonmalignant hematologic diseases is defined as the proportion of participants whose underlying disease relapses. Relapse rate of malignant and nonmalignant hematologic diseases will be provided with a 95% CI. The CI will be calculated based on the exact method for binomial distributions. Cumulative incidence rate and summary statistics will be provided.

## 7.3.8. Time to Primary Hematologic Disease Relapse

Time to primary hematologic disease relapse is defined as the interval between the date of randomization and the date of relapse. Time to the relapse will be assessed using Kaplan-Meier method. Median time to relapse and a 95% CI will be estimated. Summary statistics will be provided.

## 7.3.9. Other Efficacy Analyses

The proportion of participants with  $\geq 50\%$  reduction in daily corticosteroid dose at Day 180 will be summarized. Corticosteroid dose on study Day 1 will be defined as the starting dose as appropriate.

The proportion of participants successfully tapered off all corticosteroids at Day 180 will be summarized.

Both time to failure-free survival and average biweekly weight-standardized steroid up to Month 6 will be plotted.

## 8. PHARMACOKINETIC ANALYSES

Appendix G provides a list of planned tables and figures for the PK and PK/pharmacodynamic analyses.

## 8.1. Pharmacokinetic Analyses

In participants with full profiles (ie, in Part 1 and Part 1 expansion), the PK parameters of C<sub>max</sub>, T<sub>max</sub>, C<sub>min</sub>, AUC<sub>0-t</sub>, and Cl/F will be calculated from the blood plasma concentrations of itacitinib using standard noncompartmental (model-independent) PK methods. Pharmacokinetic calculations will be performed using commercial software such as WinNonlin<sup>®</sup> (Pharsight Corporation, Mountain View, CA).

Exposure/response analyses may be performed using model-based AUCs or using observed trough values (C<sub>min</sub>).

### 9. SAFETY AND TOLERABILITY

Appendix A provides a list of planned tables and listings.

### 9.1. General Considerations

All safety analyses will be conducted for the safety population and summarized by treatment group. Summary tables may be replaced with listings when appropriate. For instance, an AE frequency table may be replaced with a listing if it only contains a few unique PTs reported on relatively few participants.

In order to accommodate the changes proposed in Protocol Amendment 8 that resulted in discontinuation of Treatment Group C (300 mg BID) and subsequent dose reduction of ongoing participants in Treatment Group C to 400 mg QD, safety tables (specifically AEs) will be presented for the 300 mg BID group with participants who are subject to dose reduction and censored at the date of switching to the lower dose (400 mg QD). An overall summary including both dose groups (participants included before and after the dose reduction) will also be presented.

#### 9.2. Adverse Events

#### 9.2.1. Adverse Event Definitions

A TEAE is either an AE reported for the first time or worsening of a pre-existing condition after first dose of study drug until 30 days after the last dose of study drug. Analysis of AEs will be limited to TEAEs, but data listings will include all AEs, regardless of their timing in relation to study drug administration.

Adverse events will be tabulated by MedDRA PT and SOC. Severity of AEs will be described and graded using the NCI CTCAE v4.03 (NCI 2010). The CTCAE reporting guidelines and grading details are available on the Cancer Therapy Evaluation Program website.

A grading (severity) scale is provided for each AE term. If the toxicity is not included in the CTCAE v4.03, then it will be rated on a scale of 1 to 5 as follows: 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, and 5 = death due to AE. All toxicities will be graded based on the worst level reached, not the level they may have reached if they had not been treated. When the intensity of an AE changes over time for a reporting period (eg, between visits), then each change in intensity will be reported as an AE until the event resolves.

The subset of AEs considered by the investigator to be related to study drug will be considered to be treatment-related AEs. If the investigator does not specify the relationship of the AE to study drug, then the AE will be considered to be treatment-related. The incidence of AEs and treatment-related AEs will be tabulated. Serious AEs will also be tabulated.

Any missing onset date, causality, or severity must be queried for resolution. Unresolved missing values will be handled according to the following rules:

- An unresolved missing causality will be considered treatment-related.
- An unresolved missing severity will be identified as an unknown severity.

For purposes of analysis, all AEs will be considered TEAEs unless the AE can unequivocally be defined as not treatment-emergent.

## 9.2.2. **Dose-Limiting Toxicities**

Evaluation of DLTs was performed in Part 1 and in Part I expansion for the safety run-in population (first 10 participants) enrolled in Treatment Groups B and C. The toxicity of itacitinib will be monitored continuously for each treatment group using the Bayesian approach of Thall et al (1995, 1996) as extended by Thall and Sung (1998). Dose-limiting toxicities are defined in Table 5. The DLTs will be summarized on the first 28 days of study treatment.

**Table 5:** Definitions of Dose-Limiting Toxicity

| Toxicity | Definition |
|---|---|
| Nonhematologic | • Any ≥ Grade 3 nonhematologic toxicity that can be reasonably attributed to study treatment. ≥ Grade 3 nonhematologic toxicities that may be related to underlying GVHD (eg, nausea, vomiting, diarrhea, rash, dry eye) will not be considered as DLTs. |
| | • Any ≥ Grade 3 clinical chemistry laboratory abnormalities that are considered clinically significant and related to study treatment. Transient abnormal laboratory values without associated clinically significant signs and symptoms, manageable with adequate medical care, and not leading to hospitalization will not be considered as DLTs. |
| Hematologic | <ul> <li>Grade 4 neutropenia lasting more than 7 days or a ≥ 90% decrease in absolute neutrophil count from baseline that can reasonably be attributed to study treatment.</li> <li>Platelet count &lt; 10 × 10<sup>9</sup>/L related to study treatment that does not recover to at least 20 × 10<sup>9</sup>/L after 2 weeks with no requirement for platelet transfusion in the preceding 3 days.</li> </ul> |

Historical data on similar patients show a toxicity rate of 25%. The probability of toxicity for the historical data is modeled by beta distribution (Beta [25, 75]). The prior probability of toxicity for the experimental regimen is also modeled by beta distributions (Beta [0.5, 1.5]), which have the same means as the corresponding beta distributions for the historical data. Denoting the historical probability of toxicity rate by p(TOX,H), the following decision criteria will be applied:

Stop if Prob{p(TOX,H) + 
$$\delta$$
TOX < p(TOX,E)| data} > 0.95, where  $\delta$ TOX = 0

Participants from each treatment group will be monitored according to the following nonbinding stopping boundaries for toxicity in Table 6. If a boundary is reached, the sponsor and external DMC will investigate and decide on the most appropriate action.

**Table 6:** Toxicity Stopping Boundaries

| # Participants (Inclusive) | Maximum Allowable Number of Toxicities (Inclusive) |
|---|---|
| 1-2 | No limit |
| 3-4 | 3 |
| 5-6 | 4 |
| 7-9 | 5 |
| 10-11 | 6 |
| 12-14 | 7 |
| 15-17 | 8 |
| 18-19 | 9 |
| 20 | 9 |

#### 9.2.3. Adverse Event Summaries

An overall summary of AEs by treatment group will include the following:

- Number (%) of participants reporting any TEAEs
- Number (%) of participants reporting any serious TEAEs
- Number (%) of participants reporting any Grade 3 and higher TEAEs
- Number (%) of participants reporting any DLTs
- Number (%) of participants reporting any TEAEs related to itacitinib
- Number (%) of participants who temporarily interrupted itacitinib because of TEAEs
- Number (%) of participants with itacitinib dose reductions because of TEAEs
- Number (%) of participants who permanently discontinued itacitinib because of TEAEs
- Number (%) of participants reporting any TEAEs related to corticosteroid
- Number (%) of participants who temporarily interrupted corticosteroid because of TEAEs
- Number (%) of participants with corticosteroid dose reductions because of TEAEs
- Number (%) of participants who permanently discontinued corticosteroid because of TEAEs
- Number (%) of participants who had a fatal TEAE

The following summaries will be produced by MedDRA term (if 10 or fewer participants appear in a table, a listing may be appropriate):

- Number (%) of participants reporting TEAEs by SOC and PT
- Number (%) of participants reporting TEAEs by PT in decreasing order of frequency
- Number (%) of participants reporting TEAEs by SOC, PT, and maximum severity

- Number (%) of participants reporting itacitinib treatment-related TEAEs by SOC and PT
- Number (%) of participants reporting itacitinib treatment-related TEAEs by PT in decreasing order of frequency
- Number (%) of participants reporting itacitinib treatment-related, Grade 3 or higher TEAEs by SOC and PT
- Number (%) of participants reporting any Grade 3 or higher TEAEs by SOC and PT
- Number (%) of participants reporting any Grade 3 or higher TEAEs by SOC and PT in decreasing order of frequency
- Number (%) of participants reporting serious TEAEs by SOC and PT
- Number (%) of participants reporting serious TEAEs by SOC and PT in decreasing order of frequency
- Number (%) of participants reporting itacitinib treatment-related, serious TEAEs by SOC and PT
- Number (%) of participants reporting TEAEs leading to itacitinib dose interruption by SOC and PT
- Number (%) of participants reporting TEAEs leading to itacitinib dose reduction by SOC and PT
- Number (%) of participants reporting TEAEs leading to discontinuation of itacitinib by SOC and PT
- Number (%) of participants reporting corticosteroid treatment-related TEAEs by SOC and PT
- Number (%) of participants reporting corticosteroid treatment-related TEAEs by PT in decreasing order of frequency
- Number (%) of participants reporting corticosteroid treatment-related, Grade 3 or higher TEAEs by SOC and PT
- Number (%) of participants reporting corticosteroid treatment-related, serious TEAEs by SOC and PT
- Number (%) of participants reporting TEAEs leading to corticosteroid dose interruption by SOC and PT
- Number (%) of participants reporting TEAEs leading to corticosteroid dose reduction by SOC and PT
- Number (%) of participants reporting TEAEs leading to discontinuation of corticosteroids by SOC and PT
- Number (%) of participants reporting fatal TEAEs by SOC and PT

## 9.2.4. Clinically Notable Adverse Events Based on Customized MedDRA Queries

There are 9 categories of clinically notable TEAEs (ie, categories of erythropenia [anemia], neutropenia, thrombocytopenia, CMV infections, EBV infections, hyperlipidemia, QT prolongation, thromboembolic events, fungal infections) that, in particular, are of scientific and medical interest specific to itacitinib and the GVHD population. The lists of MQs are in Appendix B through Appendix F.

Within each category, the number and percentage of participants with at least 1 event occurring during treatment tabulated by MedDRA PT will be summarized. Summaries of clinically notable AEs based on customized MQs will be provided by category, PT, and the maximum severity.

## 9.3. Analyses for the Data Monitoring Committee

All safety data will be closely monitored. An external DMC will perform a full review of safety, efficacy, tolerability, and PK data. The primary purpose of the DMC is to provide a recommendation on an appropriate dose of itacitinib for Part 2.

Details of the efficacy evaluation will be included in the internal DMC charter. All safety information, including the AE data from the replaced participants, will be reviewed during this review process.

## 9.4. Clinical Laboratory Tests

Laboratory values and change from baseline values will be summarized descriptively by visit. Baseline will be determined according to Section 4.1.3. If there are multiple values that meet the criteria for baseline, additional rules may be provided after consultation with the medical monitor to delineate which value will be defined as baseline.

Laboratory data will be classified based on CTCAE grade. The incidence of abnormal laboratory values and shift tables relative to baseline will be tabulated.

## 9.5. Vital Signs

Descriptive statistics and mean change from baseline will be summarized for vital signs (ie, blood pressure, pulse, respiratory rate, and body temperature) at each assessment time. Vital sign results will be reviewed for abnormalities (see Table 7), and participants exhibiting vital sign abnormalities will be listed. A value will be considered an "alert" value if it is outside the established range and shows a > 25% change from baseline. The values for participants exhibiting alert vital sign abnormalities will be listed.

**Table 7:** Criteria for Vital Sign Abnormalities

| Parameter | High Threshold | Low Threshold |
|--------------------------|------------------|-----------------|
| Systolic blood pressure | > 155 mmHg | < 85 mmHg |
| Diastolic blood pressure | > 100 mmHg | < 40 mmHg |
| Pulse | > 100 bpm | < 45 bpm |
| Temperature | > 38°C | < 35.5°C |
| Respiratory rate | > 24 breaths/min | < 8 breaths/min |

## 9.6. Electrocardiograms

Electrocardiograms will be performed at screening and end of treatment. Electrocardiograms that are identified as abnormal and clinically meaningful compared with the screening assessment should be reported as AEs. No summary of electrocardiogram data is planned.

### 10. INTERIM ANALYSES

Preplanned analyses of safety will be provided to an independent DMC as specified in the DMC charter.

## 11. CHANGES AND MODIFICATIONS TO THE ANALYSIS PLAN

All versions of the SAP are listed in Table 8.

**Table 8:** Statistical Analysis Plan Versions

| SAP Version | Date |
|-------------|-------------|
| Original | 06 NOV 2019 |
| Amendment 1 | 03 MAR 2022 |

## 11.1. Changes to Protocol-Defined Analyses

Note that the ITT population is equivalent to the safety analysis set as defined in the Protocol.

## 11.2. Changes to the Statistical Analysis Plan

The changes reflected in this version of the SAP include the title of the study as well as Part 1 expansion details described in Protocol Amendment 7 (addition of Part 1 expansion) and Protocol Amendment 8 (closure of the BID treatment group). More specifically:

- Section 1 was updated to align with Protocol Amendment 8, which includes all details related to Part 1 expansion.
- Section 2 was updated to include all endpoints related to Part 1 expansion.
- Section 3 was updated to include the study design for Part 1 expansion.
- Section 4 was updated to include information on the corticosteroids-only group.
- Section 5 was updated to include clarifications on study populations.
- Section 6 was updated to include primary hematologic disease and transplant characteristics and to update information on exposure.
- Section 7 was updated with detailed descriptions of the efficacy endpoints to align with Protocol Amendment 8.
- Section 9 was updated to include a paragraph on the changes in Treatment Group C as outlined in Protocol Amendment 8.
- Appendix A was updated to include all tables/listings/figures intended for Part 1 expansion.

#### 12. REFERENCES

Brookmeyer R, Crowley J. A confidence interval for the median survival time. Biometrics 1982;38:29-41.

Jagasia MH, Greinix HT, Arora M, et al. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: I. The 2014 Diagnosis and Staging Working Group report. Biol Blood Marrow Transplant 2015;21:389-401.

Lee SJ, Wolff D, Kitko C, et al. Measuring therapeutic response in chronic graft-versus-host disease. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-Versus-Host Disease: IV. The 2014 Response Criteria Working Group report. Biol Blood Marrow Transplant 2015;21:984-999.

Mosteller RD. Simplified calculation of body-surface area. N Engl J Med 1987;317:1098.

National Cancer Institute. Common Terminology Criteria for Adverse Events Version 4.03. 2010.

Thall PF, Simon R, Estey EH. Bayesian sequential monitoring designs for single-arm clinical trials with multiple outcomes. Stat Med 1995;14:357-379.

Thall PF, Simon R, Estey EH. New statistical strategy for monitoring safety and efficacy in single-arm clinical trials. J Clin Oncol 1996;14:296-303.

Thall PF, Sung HG. Some extensions and applications of a Bayesian strategy for monitoring multiple outcomes in clinical trials. Stat Med 1998;17:1563-1580.

## APPENDIX A. PLANNED TABLES AND LISTINGS

This appendix provides a list of the planned tables, figures, and listings for the Clinical Study Report. Standard tables will follow the conventions in the Standard Safety Tables v1.4. In-text tables are identical in structure and content to appendix tables but follow a Rich Text Format.

Efficacy will use the safety analysis set as described in Section 5.3.

### **Tables**

| Table No. | Title | Population |
|---|---|---|
| 1.1.1.1 | Analysis Populations – Part 1 Expansion | Safety |
| 1.1.1.2 | Analysis Populations – Part 1 and Part 1 Expansion | Safety |
| 1.1.2.1 | Summary of Participant Disposition – Part 1 Expansion | Safety |
| 1.1.2.2 | Summary of Participant Disposition – Part 1 and Part 1 Expansion | Safety |
| 1.1.3.1 | Summary of Protocol Deviations – Part 1 Expansion | Safety |
| 1.1.3.2 | Summary of Protocol Deviations – Part 1 and Part 1 Expansion | Safety |
| 1.2.1.1 | Summary of Demographics – Part 1 Expansion | Safety |
| 1.2.1.2 | Summary of Demographics – Part 1 and Part 1 Expansion | Safety |
| 1.3.1.1.1 | Summary of Baseline Disease Characteristics for Cancer History – Part 1<br>Expansion | Safety |
| 1.3.1.1.2 | Summary of Baseline Disease Characteristics for Cancer History – Part 1 and Part 1 Expansion | Safety |
| 1.3.1.2.1 | Summary of Baseline Disease Characteristics for GVHD – Part 1 Expansion | Safety |
| 1.3.1.2.2 | Summary of Baseline Disease Characteristics for GVHD – Part 1 and Part 1 Expansion | Safety |
| 1.3.2.1 | Summary of Allogeneic Hematopoietic Stem Cell Transplant History – Part 1 Expansion | Safety |
| 1.3.2.2 | Summary of Allogeneic Hematopoietic Stem Cell Transplant History – Part 1 and Part 1 Expansion | Safety |
| 1.3.2.3 | Summary of Karnofsky Scale | Safety |
| 1.3.3.1 | Summary of Prior Anticancer Therapy – Part 1 Expansion | Safety |
| 1.3.3.2 | Summary of Prior Anticancer Therapy – Part 1 and Part 1 Expansion | Safety |
| 1.4.1.1 | Summary of Prior Medications – Part 1 Expansion | Safety |
| 1.4.1.2 | Summary of Prior Medications – Part 1 and Part 1 Expansion | Safety |
| 1.4.2.1 | Summary of Concomitant Medications – Part 1 Expansion | Safety |
| 1.4.2.2 | Summary of Concomitant Medications – Part 1 and Part 1 Expansion | Safety |
| 1.5.1.1 | Summary of General Medical History – Part 1 and Part 1 Expansion | Safety |
| 1.5.1.2 | Summary of Conditioning and Prophylaxis Therapy – Part 1 and Part 1 Expansion | Safety |
| 2.2.1 | Summary of Overall Response Rate at Months 3, 6, and 12 | Safety |
| 2.2.2 | Summary of Nonrelapse Mortality Rate | Safety |
| 2.2.3 | Summary of Duration of Response | Safety |
| 2.2.4 | Summary of Time to Response | Safety |
| 2.2.5 | Summary of Relapse Rate of Malignant and Nonmalignant Hematologic Diseases | Safety |
| 2.2.6 | Summary of Time to Primary Hematologic Disease Relapse | Safety |
| 2.2.7 | Summary of Overall Survival | Safety |
| 2.2.8 | Summary of Best Overall Response | Safety |
| 2.2.8.1 | Summary of Best Overall Response by GVHD Organ Involved | Safety |

| Table No. | Title | Population |
|---|---|---|
| 2.2.8.2 | Summary of Best Overall Response for Skin Sclerotic Findings Subgroup | Safety |
| 2.2.9 | Summary of Failure-Free Survival | Safety |
| 2.2.11 | Summary of Number of Participants With ≥ 50% Reduction in Daily Corticosteroid Dose at Day 180 | Safety |
| 2.2.12 | Summary of Participants Successfully Tapered Off All Corticosteroids at Day 180 | Safety |
| 2.2.13 | Summary of Number of Participants With ≥ 50% Reduction in Daily Corticosteroid Dose by (4-Week) Time Interval Up to Month 6 | Safety |
| 2.2.14 | Summary of Participants Successfully Tapered Off All Corticosteroids by (4-Week) Time Interval Up to Month 6 | Safety |
| 3.1.1 | Summary of Itacitinib Exposure, Duration of Exposure, and Dose Adjustment | Safety |
| 3.1.2 | Summary of Itacitinib Compliance | Safety |
| 3.1.3 | Summary of Corticosteroid Exposure, Duration of Exposure, and Dose Adjustment | Safety |
| 3.2.1 | Overall Summary of Treatment-Emergent Adverse Events | Safety |
| 3.2.2 | Summary of Treatment-Emergent Adverse Events by MedDRA System Organ<br>Class and Preferred Term | Safety |
| 3.2.3 | Summary of Treatment-Emergent Adverse Events by MedDRA Preferred Term in Decreasing Order of Frequency | Safety |
| 3.2.4 | Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class, Preferred Term, and Maximum Severity | Safety |
| 3.2.5 | Summary of Itacitinib Treatment-Related, Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term | Safety |
| 3.2.6 | Summary of Itacitinib Treatment-Related, Treatment-Emergent Adverse Events by MedDRA Preferred Term in Decreasing Order of Frequency | Safety |
| 3.2.7 | Summary of Itacitinib Treatment-Related, Grade 3 or Higher Treatment-Emergent Adverse Events by MedDRA System Organ Class, and Preferred Term | Safety |
| 3.2.8 | Summary of Grade 3 or Higher Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term | Safety |
| 3.2.9 | Summary of Grade 3 or Higher Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term in Decreasing Order of Frequency | Safety |
| 3.2.10 | Summary of Serious Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term | Safety |
| 3.2.11 | Summary of Serious Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term in Decreasing Order of Frequency | Safety |
| 3.2.12 | Summary of Itacitinib Treatment-Related, Serious Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term | Safety |
| 3.2.13 | Summary of Treatment-Emergent Adverse Events Leading to Itacitinib Dose<br>Interruption by MedDRA System Organ Class and Preferred Term | Safety |
| 3.2.14 | Summary of Treatment-Emergent Adverse Events Leading to Itacitinib Dose<br>Reduction by MedDRA System Organ Class and Preferred Term | Safety |
| 3.2.15 | Summary of Treatment-Emergent Adverse Events Leading to Discontinuation of Itacitinib by MedDRA System Organ Class and Preferred Term | Safety |
| 3.2.16 | Summary of Corticosteroid Treatment-Related, Treatment-Emergent Adverse<br>Events by MedDRA System Organ Class and Preferred Term | Safety |
| 3.2.17 | Summary of Corticosteroid Treatment-Related, Treatment-Emergent Adverse Events by MedDRA Preferred Term in Decreasing Order of Frequency | Safety |
| 3.2.18 | Summary of Corticosteroid Treatment-Related, Serious Treatment-Emergent<br>Adverse Events by MedDRA System Organ Class and Preferred Term | Safety |

| Table No. | Title | Population |
|---|---|---|
| 3.2.19 | Summary of Treatment-Emergent Adverse Events Leading to Corticosteroid Dose Interruption by MedDRA System Organ Class and Preferred Term | Safety |
| 3.2.20 | Summary of Treatment-Emergent Adverse Events Leading to Corticosteroid Dose<br>Reduction by MedDRA System Organ Class and Preferred Term | Safety |
| 3.2.21 | Summary of Treatment-Emergent Adverse Events Leading to Discontinuation of Corticosteroid by MedDRA System Organ Class and Preferred Term | Safety |
| 3.2.22 | Summary of Treatment-Emergent Adverse Events With a Fatal Outcome by MedDRA System Organ Class and Preferred Term | Safety |
| 3.2.23 | Overall Summary of Treatment-Emergent Clinically Notable Hematologic Events by Customized MQs | Safety |
| 3.2.24 | Summary of Clinically Notable Treatment-Emergent Hematologic Events by Customized MQs, Preferred Term, and Maximum Severity | Safety |
| 3.2.25 | Overall Summary of Treatment-Emergent CMV Infection Events by Customized MedDRA Queries | Safety |
| 3.2.26 | Summary of Treatment-Emergent CMV Infection Events by Customized MedDRA Queries, Preferred Term, and Maximum Severity | Safety |
| 3.2.27 | Overall Summary of Treatment-Emergent EBV Infection Events by Customized MedDRA Queries | Safety |
| 3.2.28 | Summary of Treatment-Emergent EBV Infection Events by Customized MedDRA Queries, Preferred Term, and Maximum Severity | Safety |
| 3.2.29 | Overall Summary of Treatment-Emergent Hyperlipidemia Events by Customized MedDRA Queries | Safety |
| 3.2.30 | Summary of Treatment-Emergent Hyperlipidemia Events by Customized MedDRA Queries, Preferred Term, and Maximum Severity | Safety |
| 3.2.31 | Summary of Grade 3 or Higher Treatment-Emergent Infections by MedDRA System Organ Class and Preferred Term | Safety |
| 3.2.32 | Summary of Treatment-Emergent CMV Infection Events by MedDRA System Organ Class and Preferred Term | Safety |
| 3.2.33 | Summary of Treatment-Emergent QT Prolongation Events by Customized MedDRA Queries, Preferred Term, and Maximum Severity | Safety |
| 3.2.34 | Overall Summary of Treatment-Emergent Thromboembolic Events by Customized MedDRA Queries | Safety |
| 3.2.35 | Summary of Treatment-Emergent Thromboembolic Events by Customized MedDRA Queries, Preferred Term, and Maximum Severity | Safety |
| 3.2.36 | Overall Summary of Treatment-Emergent Fungal Infection Events (MedDRA High<br>Level Group Term) by Customized MedDRA Queries | Safety |
| 3.2.37 | Summary of Treatment-Emergent Fungal Infection Events (MedDRA High Level Group Term) by Customized MedDRA Queries, Preferred Term, and Maximum Severity | Safety |
| 3.3.1.1 | Summary of Laboratory Values – Hematology | Safety |
| 3.3.1.2 | Shift Summary of Hematology Laboratory Values in CTCAE Grade – to the Worst Abnormal Value | Safety |
| 3.3.2.1 | Summary of Laboratory Values – Chemistry | Safety |
| 3.3.2.2 | Shift Summary of Chemistry Laboratory Values in CTCAE Grade – to the Worst Abnormal Value | Safety |
| 3.3.3.1 | Summary of Laboratory Values - Coagulation | Safety |
| 3.4.1 | Summary of Systolic Blood Pressure | Safety |
| 3.4.2 | Summary of Diastolic Blood Pressure | Safety |

| Table No. | Title | Population |
|-----------|-----------------------------|------------|
| 3.4.3 | Summary of Pulse | Safety |
| 3.4.4 | Summary of Respiratory Rate | Safety |
| 3.4.5 | Summary of Body Temperature | Safety |
| 3.4.6 | Summary of Body Weight | Safety |

## Figures

| Figure No. | Title |
|------------|------------------------------------------------------------|
| 4.2.1 | Kaplan-Meier Plot of Time to Failure-Free Survival |
| 4.3.1 | Average Biweekly Weight-Standardized Steroid Up to Month 6 |

## Listings

| Listing No. | Title |
|---|---|
| 2.1.1 | Participant Enrollment and Disposition Status |
| 2.4.7 | Posttherapy Medications |
| 2.6.8 | Deaths |
| 2.7.7 | Adverse Events Leading to Interruption, Reduction, or Discontinuation of Itacitinib |
| 99.2.1 | Protocol Deviations by Deviation Coded Term |

## APPENDIX B. CLINICALLY NOTABLE HEMATOLOGIC EVENTS

This appendix provides a list of 3 categories of clinically notable treatment-emergent hematologic events based on customized MQs.

| <b>Adverse Event Category</b> | Preferred Term | Code |
|---|---|---|
| Anemia | Anaemia macrocytic | 10002064 |
| | Aplasia pure red cell | 10002965 |
| | Aplastic anaemia | 10002967 |
| | Erythroblast count decreased | 10058505 |
| | Erythropenia | 10015287 |
| | Hypoplastic anaemia | 10021074 |
| | Microcytic anaemia | 10027538 |
| | Red blood cell count decreased | 10038153 |
| | Anaemia | 10002034 |
| | Haematocrit decreased | 10018838 |
| | Haemoglobin decreased | 10018884 |
| | Leukoerythroblastic anaemia | 10053199 |
| | Normochromic normocytic anaemia | 10029783 |
| Neutropenia | Agranulocytosis | 10001507 |
| | Band neutrophil count decreased | 10057950 |
| | Febrile neutropenia | 10016288 |
| | Granulocyte count decreased | 10018681 |
| | Granulocytopenia | 10018687 |
| | Neutropenia | 10029354 |
| | Neutropenic infection | 10059482 |
| | Neutropenic sepsis | 10049151 |
| | Neutrophil count decreased | 10029366 |
| Thrombocytopenia | Acquired amegakaryocytic thrombocytopenia | 10076747 |
| | Platelet count decreased | 10035528 |
| | Thrombocytopenia | 10043554 |
| | Plateletcrit decreased | 10064784 |

## APPENDIX C. HEMATOLOGIC INFECTION EVENTS

| <b>Adverse Event Group</b> | Preferred Term | Code |
|---|---|---|
| EBV infections | Epstein-Barr virus positive mucocutaneous ulcer | 10079386 |
| | Epstein-Barr viraemia | 10065110 |
| | Epstein-Barr virus associated lymphoma | 10071441 |
| | Epstein-Barr virus associated lymphoproliferative disorder | 10068349 |
| | Epstein-Barr virus infection | 10015108 |
| | Hepatitis infectious mononucleosis | 10019781 |
| | Infectious mononucleosis | 10021914 |
| | Oral hairy leukoplakia | 10030979 |
| | Post transplant lymphoproliferative disorder | 10051358 |
| | X-linked lymphoproliferative syndrome | 10068348 |
| | Epstein-Barr virus test positive | 10064545 |
| | Epstein-Barr virus antibody positive | 10052324 |
| Cytomegaloviral infections | Congenital cytomegalovirus infection | 10010430 |
| | Cytomegalovirus chorioretinitis | 10048843 |
| | Cytomegalovirus colitis | 10048983 |
| | Cytomegalovirus duodenitis | 10049014 |
| | Cytomegalovirus enteritis | 10049074 |
| | Cytomegalovirus enterocolitis | 10049015 |
| | Cytomegalovirus gastritis | 10049016 |
| | Cytomegalovirus gastroenteritis | 10051349 |
| | Cytomegalovirus gastrointestinal infection | 10052817 |
| | Cytomegalovirus gastrointestinal ulcer | 10075619 |
| | Cytomegalovirus hepatitis | 10011830 |
| | Cytomegalovirus infection | 10011831 |
| | Cytomegalovirus mononucleosis | 10011834 |
| | Cytomegalovirus mucocutaneous ulcer | 10065036 |
| | Cytomegalovirus myelomeningoradiculitis | 10065621 |
| | Cytomegalovirus myocarditis | 10056261 |
| | Cytomegalovirus nephritis | 10079095 |
| | Cytomegalovirus oesophagitis | 10049018 |
| | Cytomegalovirus pancreatitis | 10049566 |
| | Cytomegalovirus pericarditis | 10056721 |
| | Cytomegalovirus syndrome | 10056262 |
| | Cytomegalovirus urinary tract infection | 10051350 |
| | Cytomegalovirus viraemia | 10058854 |
| | Encephalitis cytomegalovirus | 10014586 |
| | Disseminated cytomegaloviral infection | 10049075 |
| | Pneumonia cytomegaloviral | 10035676 |
| | Cytomegalovirus test positive | 10051620 |

## APPENDIX D. HYPERLIPIDEMIA EVENTS

| Preferred Term | Code | Level | Scope | Category | Weight | Status | Addition<br>Version | Last<br>Modified<br>Version |
|---|---|---|---|---|---|---|---|---|
| Acquired lipoatrophic diabetes | 10073667 | PT | Narrow | A | 0 | Active | 16.1 | 16.1 |
| Acquired mixed hyperlipidaemia | 10071236 | PT | Narrow | A | 0 | Active | 18.0 | 18.0 |
| Apolipoprotein<br>B/Apolipoprotein A-1 ratio<br>increased | 10065516 | PT | Narrow | A | 0 | Active | 13.0 | 13.0 |
| Autoimmune<br>hyperlipidaemia | 10071577 | PT | Narrow | A | 0 | Active | 14.1 | 14.1 |
| Blood cholesterol abnormal | 10005423 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| Blood cholesterol esterase increased | 10071304 | PT | Narrow | A | 0 | Active | 14.1 | 14.1 |
| Blood cholesterol increased | 10005425 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| Blood triglycerides abnormal | 10005837 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| Blood triglycerides increased | 10005839 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| Diabetic dyslipidaemia | 10070901 | PT | Narrow | A | 0 | Active | 14.0 | 14.0 |
| Dyslipidaemia | 10058108 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| High density lipoprotein abnormal | 10020051 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| High density lipoprotein decreased | 10020060 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| Hypercholesterolaemia | 10020603 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| Hyperlipidaemia | 10062060 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| Hypertriglyceridaemia | 10020869 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| Hypo HDL cholesterolaemia | 10068961 | PT | Narrow | A | 0 | Active | 12.0 | 12.0 |
| Intermediate density lipoprotein increased | 10064236 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| LDL/HDL ratio increased | 10049030 | PT | Narrow | A | 0 | Active | 13.0 | 13.0 |
| Lipids abnormal | 10024588 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| Lipids increased | 10024592 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| Lipoprotein (a) abnormal | 10054023 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| Lipoprotein (a) increased | 10054009 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| Lipoprotein abnormal | 10081355 | PT | Narrow | A | 0 | Active | 21.1 | 21.1 |
| Lipoprotein increased | 10081354 | PT | Narrow | A | 0 | Active | 21.1 | 21.1 |
| Low density lipoprotein abnormal | 10024901 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| Low density lipoprotein increased | 10024910 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |

| Preferred Term | Code | Level | Scope | Category | Weight | Status | Addition<br>Version | Last<br>Modified<br>Version |
|---|---|---|---|---|---|---|---|---|
| Non-high-density lipoprotein cholesterol increased | 10063967 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| Remnant-like lipoprotein particles increased | 10073041 | PT | Narrow | A | 0 | Active | 16.0 | 16.0 |
| Total cholesterol/HDL ratio abnormal | 10058633 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| Total cholesterol/HDL ratio increased | 10058630 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| Very low density lipoprotein abnormal | 10047352 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |
| Very low density lipoprotein increased | 10047361 | PT | Narrow | A | 0 | Active | 8.1 | 8.1 |

## APPENDIX E. QT PROLONGATION EVENTS

| Preferred Term | Code | Level | Scope | Category | Weight | Status | Addition<br>Version | Last<br>Modified<br>Version |
|---|---|---|---|---|---|---|---|---|
| Electrocardiogram<br>QT interval abnormal | 10063748 | PT | Narrow | A | 0 | Active | 7.1 | 7.1 |
| Electrocardiogram<br>QT prolonged | 10014387 | PT | Narrow | A | 0 | Active | 7.1 | 7.1 |
| Long QT syndrome | 10024803 | PT | Narrow | A | 0 | Active | 7.1 | 7.1 |
| Long QT syndrome congenital | 10057926 | PT | Narrow | A | 0 | Active | 7.1 | 7.1 |
| Torsade de pointes | 10044066 | PT | Narrow | A | 0 | Active | 7.1 | 7.1 |
| Ventricular tachycardia | 10047302 | PT | Narrow | A | 0 | Active | 7.1 | 7.1 |

## APPENDIX F. THROMBOEMBOLIC EVENTS

| | | | | | | | | Addition | Last<br>Modified |
|---|---|---|---|---|---|---|---|---|---|
| Group | Preferred Term | Code | Level | Scope | Category | Weight | Status | Version | Version |
| Arterial | Acute aortic syndrome | 10074337 | PT | Narrow | A | 0 | Active | 17.0 | 17.0 |
| | Acute myocardial infarction | 10000891 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Amaurosis | 10001902 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Amaurosis fugax | 10001903 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Angioplasty | 10002475 | PT | Narrow | A | 0 | Active | 16.0 | 16.0 |
| | Aortic bypass | 10057617 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Aortic embolus | 10002897 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Aortic surgery | 10061651 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Aortic thrombosis | 10002910 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Aortogram abnormal | 10057794 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Arterectomy | 10071026 | PT | Narrow | A | 0 | Active | 14.0 | 14.0 |
| | Arterectomy with graft replacement | 10003140 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Arterial angioplasty | 10081731 | PT | Narrow | A | 0 | Active | 21.1 | 21.1 |
| | Arterial bypass occlusion | 10077766 | PT | Narrow | A | 0 | Active | 19.0 | 19.0 |
| | Arterial bypass operation | 10056418 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Arterial bypass thrombosis | 10077765 | PT | Narrow | A | 0 | Active | 19.0 | 19.0 |
| | Arterial graft | 10061655 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Arterial occlusive disease | 10062599 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Arterial stent insertion | 10061657 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Arterial therapeutic procedure | 10052949 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Arterial thrombosis | 10003178 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Arteriogram abnormal | 10061659 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Arteriogram carotid abnormal | 10003195 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Arteriotomy | 10078636 | PT | Narrow | A | 0 | Active | 19.1 | 19.1 |
| | Atherectomy | 10063025 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Atherosclerotic plaque rupture | 10076604 | PT | Narrow | A | 0 | Active | 18.1 | 18.1 |
| | Atrial appendage closure | 10079735 | PT | Narrow | A | 0 | Active | 20.1 | 20.1 |
| | Atrial appendage resection | 10080843 | PT | Narrow | A | 0 | Active | 21.0 | 21.0 |
| | Basal ganglia infarction | 10069020 | PT | Narrow | A | 0 | Active | 12.0 | 12.0 |
| | Basilar artery occlusion | 10048963 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Basilar artery thrombosis | 10063093 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Blindness transient | 10005184 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Brachiocephalic artery occlusion | 10069694 | PT | Narrow | A | 0 | Active | 13.0 | 13.0 |
| | Capsular warning syndrome | 10067744 | PT | Narrow | A | 0 | Active | 10.1 | 10.1 |
| | Carotid angioplasty | 10071260 | PT | Narrow | A | 0 | Active | 14.1 | 14.1 |
| | Carotid arterial embolus | 10007684 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Carotid artery bypass | 10053003 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Carotid artery occlusion | 10048964 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Carotid artery stent insertion | 10066102 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Carotid artery thrombosis | 10007688 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Carotid endarterectomy | 10007692 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Cerebellar artery occlusion | 10053633 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Cerebellar artery thrombosis | 10008023 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| Arterial | Cerebral artery embolism | 10008088 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Cerebral artery occlusion | 10008089 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |

| Group | Preferred Term | Code | Level | Scope | Category | Weight | Status | Addition<br>Version | Last<br>Modified<br>Version |
|---|---|---|---|---|---|---|---|---|---|
| | Cerebral artery stent insertion | 10081893 | PT | Narrow | A | 0 | Active | 22.0 | 22.0 |
| | Cerebral artery thrombosis | 10008092 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Cerebral hypoperfusion | 10065384 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Cerebrovascular insufficiency | 10058842 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Cerebrovascular stenosis | 10061751 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Coeliac artery occlusion | 10069696 | PT | Narrow | A | 0 | Active | 13.0 | 13.0 |
| | Coronary angioplasty | 10050329 | PT | Narrow | A | 0 | Active | 16.0 | 16.0 |
| | Coronary arterial stent insertion | 10052086 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Coronary artery bypass | 10011077 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Coronary artery embolism | 10011084 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Coronary artery occlusion | 10011086 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Coronary artery reocclusion | 10053261 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Coronary artery surgery | 10011090 | PT | Narrow | A | 0 | Active | 10.0 | 20.1 |
| | Coronary artery thrombosis | 10011091 | PT | Narrow | A | 0 | Active | 16.0 | 16.0 |
| | Coronary endarterectomy | 10011101 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Coronary revascularisation | 10049887 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Coronary vascular graft occlusion | 10075162 | PT | Narrow | A | 0 | Active | 17.1 | 17.1 |
| | Embolia cutis medicamentosa | 10058729 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Embolism arterial | 10014513 | PT | Narrow | A | 0 | Active | 10.0 | 13.1 |
| | Endarterectomy | 10014648 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Femoral artery embolism | 10068365 | PT | Narrow | A | 0 | Active | 11.1 | 11.1 |
| | Hepatic artery embolism | 10019635 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Hepatic artery occlusion | 10051991 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Hepatic artery thrombosis | 10019636 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Hypothenar hammer syndrome | 10063518 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Iliac artery embolism | 10021338 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Iliac artery occlusion | 10064601 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Intra-aortic balloon placement | 10052989 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Intraoperative cerebral artery occlusion | 10056382 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Ischaemic cerebral infarction | 10060840 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Ischaemic stroke | 10061256 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Lacunar infarction | 10051078 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Leriche syndrome | 10024242 | PT | Narrow | A | 0 | Active | 13.1 | 13.1 |
| | Mesenteric arterial occlusion | 10027394 | PT | Narrow | A | 0 | Active | 17.0 | 17.0 |
| | Mesenteric arteriosclerosis | 10065560 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Mesenteric artery embolism | 10027395 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Mesenteric artery stenosis | 10027396 | | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Mesenteric artery stent insertion | 10071261 | PT | Narrow | A | 0 | Active | 14.1 | 14.1 |
| | Mesenteric artery thrombosis | 10027397 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Myocardial infarction | 10028596 | | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Myocardial necrosis | 10028602 | PT | Narrow | A | 0 | Active | 10.0 | 17.0 |
| | Ophthalmic artery thrombosis | 10081144 | PT | Narrow | A | 0 | Active | 21.1 | 21.1 |
| | Papillary muscle infarction | 10033697 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Penile artery occlusion | 10068035 | PT | Narrow | A | 0 | Active | 11.0 | 11.0 |
| Arterial | Percutaneous coronary intervention | 10065608 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| 711101101 | Peripheral arterial occlusive disease | 10062585 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |

| Group | Preferred Term | Code | Level | Scope | Category | Weight | Status | Addition<br>Version | Last<br>Modified<br>Version |
|---|---|---|---|---|---|---|---|---|---|
| • | Peripheral arterial reocclusion | 10069379 | PT | Narrow | A | 0 | Active | 12.1 | 12.1 |
| | Peripheral artery angioplasty | 10057518 | | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Peripheral artery bypass | 10072561 | PT | Narrow | A | 0 | Active | 15.1 | 15.1 |
| | Peripheral artery occlusion | 10057525 | PT | Narrow | A | 0 | Active | 10.0 | 19.0 |
| | Peripheral artery stent insertion | 10072562 | PT | Narrow | A | 0 | Active | 15.1 | 15.1 |
| | Peripheral artery surgery | 10082470 | PT | Narrow | A | 0 | Active | 22.0 | 22.0 |
| | Peripheral artery thrombosis | 10072564 | PT | Narrow | A | 0 | Active | 15.1 | 15.1 |
| | Peripheral embolism | 10061340 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Peripheral endarterectomy | 10072560 | PT | Narrow | A | 0 | Active | 15.1 | 15.1 |
| | Popliteal artery entrapment syndrome | 10071642 | PT | Narrow | A | 0 | Active | 14.1 | 14.1 |
| | Post procedural myocardial infarction | 10066592 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Postinfarction angina | 10058144 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Precerebral artery occlusion | 10036511 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Precerebral artery thrombosis | 10074717 | PT | Narrow | A | 0 | Active | 17.0 | 17.0 |
| | Profundaplasty | 10078867 | PT | Narrow | A | 0 | Active | 20.0 | 20.0 |
| | Pulmonary artery occlusion | 10078201 | PT | Narrow | A | 0 | Active | 19.1 | 19.1 |
| | Pulmonary artery therapeutic procedure | 10063731 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Pulmonary artery thrombosis | 10037340 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Pulmonary endarterectomy | 10072893 | PT | Narrow | A | 0 | Active | 16.0 | 16.0 |
| | Pulmonary tumour thrombotic microangiopathy | 10079988 | PT | Narrow | A | 0 | Active | 20.1 | 20.1 |
| | Renal artery angioplasty | 10057493 | PT | Narrow | A | 0 | Active | 15.1 | 15.1 |
| | Renal artery occlusion | 10048988 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Renal artery thrombosis | 10038380 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Renal embolism | 10063544 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Retinal artery embolism | 10038826 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Retinal artery occlusion | 10038827 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Retinal artery thrombosis | 10038831 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Silent myocardial infarction | 10049768 | PT | Narrow | A | 0 | Active | 12.1 | 12.1 |
| | Spinal artery embolism | 10049440 | | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Spinal artery thrombosis | 10071316 | PT | Narrow | A | 0 | Active | 14.1 | 14.1 |
| | Splenic artery thrombosis | 10074600 | PT | Narrow | A | 0 | Active | 17.0 | 17.0 |
| | Splenic embolism | 10068677 | PT | Narrow | A | 0 | Active | 11.1 | 11.1 |
| | Stress cardiomyopathy | 10066286 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Subclavian artery embolism | 10042332 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Subclavian artery occlusion | 10069695 | PT | Narrow | A | 0 | Active | 13.0 | 13.0 |
| | Subclavian artery thrombosis | 10042334 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Thromboembolectomy | 10064958 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Thrombotic microangiopathy | 10043645 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Thrombotic thrombocytopenic purpura | 10043648 | | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Transient ischaemic attack | 10044390 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Truncus coeliacus thrombosis | 10062363 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Vascular pseudoaneurysm thrombosis | 10078269 | PT | Narrow | A | 0 | Active | 19.1 | 19.1 |

| Group | Preferred Term | Code | Level | Scope | Category | Weight | Status | Addition<br>Version | Last<br>Modified<br>Version |
|---|---|---|---|---|---|---|---|---|---|
| Arterial | Vertebral artery occlusion | 10048965 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Vertebral artery thrombosis | 10057777 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Visual acuity reduced transiently | 10047532 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| Venous | Axillary vein thrombosis | 10003880 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Brachiocephalic vein occlusion | 10076837 | PT | Narrow | A | 0 | Active | 18.1 | 18.1 |
| | Brachiocephalic vein thrombosis | 10063363 | PT | Narrow | A | 0 | Active | 10.0 | 19.1 |
| | Budd-Chiari syndrome | 10006537 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Catheterisation venous | 10052698 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Cavernous sinus thrombosis | 10007830 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Central venous catheterisation | 10053377 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Cerebral venous sinus thrombosis | 10083037 | PT | Narrow | A | 0 | Active | 22.1 | 22.1 |
| | Cerebral venous thrombosis | 10008138 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Compression garment application | 10079209 | PT | Narrow | A | 0 | Active | 20.0 | 20.0 |
| | Deep vein thrombosis | 10051055 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Deep vein thrombosis postoperative | 10066881 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Embolism venous | 10014522 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Hepatic vein embolism | 10078810 | PT | Narrow | A | 0 | Active | 20.0 | 20.0 |
| | Hepatic vein occlusion | 10058991 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Hepatic vein thrombosis | 10019713 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Homans' sign positive | 10051031 | PT | Narrow | A | 0 | Active | 14.0 | 14.0 |
| | Iliac vein occlusion | 10058992 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Inferior vena cava syndrome | 10070911 | PT | Narrow | A | 0 | Active | 14.0 | 14.0 |
| | Inferior vena caval occlusion | 10058987 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Jugular vein embolism | 10081850 | PT | Narrow | A | 0 | Active | 22.0 | 22.0 |
| | Jugular vein occlusion | 10076835 | PT | Narrow | A | 0 | Active | 18.1 | 18.1 |
| | Jugular vein thrombosis | 10023237 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Mahler sign | 10075428 | PT | Narrow | A | 0 | Active | 17.1 | 17.1 |
| | May-Thurner syndrome | 10069727 | PT | Narrow | A | 0 | Active | 13.0 | 13.0 |
| | Mesenteric vein thrombosis | 10027402 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Mesenteric venous occlusion | 10027403 | PT | Narrow | A | 0 | Active | 17.0 | 17.0 |
| | Obstetrical pulmonary embolism | 10029925 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Obstructive shock | 10073708 | PT | Narrow | A | 0 | Active | 16.1 | 16.1 |
| | Ophthalmic vein thrombosis | 10074349 | PT | Narrow | A | 0 | Active | 17.0 | 17.0 |
| | Ovarian vein thrombosis | 10072059 | PT | Narrow | A | 0 | Active | 15.0 | 15.0 |
| | Paget-Schroetter syndrome | 10050216 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Pelvic venous thrombosis | 10034272 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Penile vein thrombosis | 10034324 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Peripheral vein occlusion | 10083103 | PT | Narrow | A | 0 | Active | 22.1 | 22.1 |
| | Peripheral vein thrombus extension | 10082853 | PT | Narrow | A | 0 | Active | 22.1 | 22.1 |
| | Phlebectomy | 10048874 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Portal vein cavernous transformation | 10073979 | PT | Narrow | A | 0 | Active | 16.1 | 16.1 |
| | Portal vein embolism | 10082030 | PT | Narrow | A | 0 | Active | 22.0 | 22.0 |
| | Portal vein occlusion | 10058989 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Portal vein thrombosis | 10036206 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Portosplenomesenteric venous thrombosis | 10077623 | PT | Narrow | A | 0 | Active | 19.0 | 19.0 |

| Crown | Preferred Term | Code | Lovel | Saama | Catagomy | Waight | Status | Addition<br>Version | Last<br>Modified<br>Version |
|---|---|---|---|---|---|---|---|---|---|
| Group | Post procedural pulmonary | 10063909 | Level<br>PT | Scope<br>Narrow | Category | Weight 0 | Status<br>Active | 10.0 | 10.0 |
| | embolism | 10003909 | PI | Narrow | A | 0 | Active | 10.0 | 10.0 |
| Venous | Post thrombotic syndrome | 10048591 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Postoperative thrombosis | 10050902 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Postpartum venous thrombosis | 10036300 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Pulmonary embolism | 10037377 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Pulmonary infarction | 10037410 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Pulmonary microemboli | 10037421 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Pulmonary thrombosis | 10037427 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Pulmonary vein occlusion | 10068690 | PT | Narrow | A | 0 | Active | 11.1 | 11.1 |
| | Pulmonary veno-occlusive disease | 10037458 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Pulmonary venous thrombosis | 10037459 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Renal vein embolism | 10037439 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Renal vein occlusion | 10056293 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Renal vein declusion Renal vein thrombosis | 10038548 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Retinal vein occlusion | 10038348 | PT | Narrow | | 0 | Active | 10.0 | 10.0 |
| | Retinal vein occusion Retinal vein thrombosis | 10038907 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | | | PT | | A | 0 | Active | 22.1 | |
| | Septic pulmonary embolism | 10083093 | | Narrow | A | | | | 22.1 |
| | SI QIII TIII pattern | 10068479 | PT | Narrow | A | 0 | Active | 11.1 | 11.1 |
| | Splenic vein occlusion | 10068122 | PT | Narrow | A | 0 | Active | 11.0 | 11.0 |
| | Splenic vein thrombosis | 10041659 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Subclavian vein occlusion | 10079164 | PT | Narrow | A | 0 | Active | 20.0 | 20.0 |
| | Subclavian vein thrombosis | 10049446 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Superior sagittal sinus thrombosis | 10042567 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Superior vena cava occlusion | 10058988 | PT | Narrow | A | 0 | Active | 10.0 | 17.0 |
| | Superior vena cava syndrome | 10042569 | PT | Narrow | A | 0 | Active | 10.0 | 14.0 |
| | Thrombophlebitis | 10043570 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Thrombophlebitis migrans | 10043581 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Thrombophlebitis neonatal | 10043586 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Thrombophlebitis superficial | 10043595 | PT | Narrow | A | 0 | Active | 14.1 | 14.1 |
| | Thrombosed varicose vein | 10043605 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Thrombosis corpora cavernosa | 10067270 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Transverse sinus thrombosis | 10044457 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Vena cava embolism | 10047193 | | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Vena cava filter insertion | 10048932 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Vena cava filter removal | 10074397 | PT | Narrow | A | 0 | Active | 17.0 | 17.0 |
| | Vena cava thrombosis | 10047195 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Venogram abnormal | 10047209 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Venoocclusive disease | 10062173 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Venoocclusive liver disease | 10047216 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Venous angioplasty | 10077826 | PT | Narrow | A | 0 | Active | 19.0 | 19.0 |
| | Venous occlusion | 10058990 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Venous operation | 10062175 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Venous recanalisation | 10068605 | PT | Narrow | A | 0 | Active | 11.1 | 11.1 |
| | Venous repair | 10052964 | PT | Narrow | A | 0 | Active | 17.1 | 17.1 |
| | Venous stent insertion | 10063389 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Venous thrombosis | 10047249 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |

| Group | Preferred Term | Code | Level | Scope | Category | Weight | Status | Addition<br>Version | Last<br>Modified<br>Version |
|---|---|---|---|---|---|---|---|---|---|
| | Venous thrombosis in pregnancy | 10067030 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| Venous | Venous thrombosis limb | 10061408 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Venous thrombosis neonatal | 10064602 | PT | Narrow | A | 0 | Active | 10.0 | 10.0 |
| | Visceral venous thrombosis | 10077829 | PT | Narrow | A | 0 | Active | 19.0 | 19.0 |

# APPENDIX G. PLANNED TABLES AND FIGURES FOR PHARMACOKINETIC AND PHARMACOKINETIC/PHARMACODYNAMIC ANALYSIS

#### **Tables**

| Table No. | Title |
|---|---|
| Table 1 | Summarization of the Pharmacokinetic Parameters by Dose at Day 1 |
| Table 2 | Summarization of the Pharmacokinetic Parameters by Dose at Day 7 |
| Table 3 | Summarization of the Pharmacokinetic Parameters by Dose at Day 28 |

**Figures** 

| Figure No. | Title |
|---|---|
| Figure 1 | Mean (± SE) Concentration-Time Profiles by Dose at Day 1 |
| Figure 2 | Boxplots of C <sub>max</sub> , C <sub>min</sub> , and AUC on Day 7 by NRM at 6 Months |
| Figure 3 | Boxplots of C <sub>max</sub> , C <sub>min</sub> , and AUC on Day 7 by Overall Response at 6 Months |
| Figure 4 | Boxplots of C <sub>max</sub> , C <sub>min</sub> , and AUC on Day 7 by Chronic GVHD Grading at 6 Months |
| Figure 5 | Boxplots of C <sub>max</sub> , C <sub>min</sub> , and AUC on Day 7 by Chronic GVHD Liver Staging at Day 7 |
| Figure 6 | Boxplots of C <sub>max</sub> , C <sub>min</sub> , and AUC on Day 28 by Chronic GVHD Liver Staging at Day 28 |
| Figure 7 | Boxplots of C <sub>max</sub> , C <sub>min</sub> , and AUC on Day 7 by Chronic GVHD GI Staging at Day 7 |
| Figure 8 | Boxplots of C <sub>max</sub> , C <sub>min</sub> , and AUC on Day 28 by Chronic GVHD GI Staging at Day 28 |

Pharmacokinetic tables and/or figures may be modified or additional PK tables and/or figures may be created as needed based on study findings. For example, plots may be modified to indicate participants taking potent CYP3A4 inhibitors and those who are not, or plots may be modified to highlight a participant who had a particular safety finding.